CLINICAL TRIAL: NCT01439243
Title: Randomized, Open-Label, 2-Way Crossover, Bioequivalence Study of Donepezil (Test) 10 mg Tablet and Aricept® (Reference) Following a 10 mg Dose in Healthy Subjects Under Fed Conditions
Brief Title: Donepezil 10 mg Tablets Under Fed Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Teva Pharmaceuticals USA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: 70186
Record Dates: First submitted 2011-09-20; First posted 2011-09-23 (Estimated); Last update posted 2011-09-23 (Estimated); Status verified 2011-09

CONDITIONS: Healthy
Keywords: Bioequivalence; Healthy Subjects; Donepezil
MeSH Terms: interventions — Donepezil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Investigational Test Product (Experimental): Donepezil 10 mg Tablets
  Interventions: Drug: Donepezil
- Reference Listed Drug (Active Comparator): Aricept® 10 mg Tablets
  Interventions: Drug: Aricept®

INTERVENTIONS:
Drug: Donepezil — 10 mg Tablet
  Arms: Investigational Test Product
Drug: Aricept® — 10 mg Tablet
  Other Names: Donepezil (generic name)
  Arms: Reference Listed Drug

SUMMARY:
The objective of this study was to compare the rate and extent of absorption of donepezil 10 mg tablet (test) versus Aricept® (reference), administered as 1 x 10 mg tablet under fed conditions.

DETAILED DESCRIPTION:
Criteria for Evaluation: FDA Bioequivalence Criteria

Statistical Method: FDA Bioequivalence Statistical Methods

ELIGIBILITY:
Inclusion Criteria:

* Male or female, non-smoker, > 18 and < 55 years of age.
* Capable of consent.
* BMI > 19.0 and < 27.0.
* Good state of health (no clinically significant deviations from normal clinical results and laboratory test findings).

Exclusion Criteria:

* Absence of any inclusion criteria.
* Clinically significant illnesses (including hyperglycemia, any form of diabetes or glucose intolerance, congestive heart failure, hepatitis, hypotensive episodes) or surgery within 8 weeks prior to dosing.
* All clinically significant abnormality or abnormal laboratory test results found during medical screening.
* Any reason which, in the opinion of the Medical Sub-Investigator, would prevent the subject from participating in the study.
* Positive test for hepatitis B. hepatitis C, or HIV at screening.
* ECG abnormalities (clinically significant) or vital sign abnormalities (systolic blood pressure lower than 95 or over 140 mmHg, diastolic blood pressure lower than 50 or over 90 mmHg, or heart rate less than 50 or over 100 bpm) at screening.
* History of significant alcohol abuse or drug abuse within 1 year prior to the screening visit.
* Regular use of alcohol within 12 months prior to the screening visit (more than 14 units of alcohol per week [1 unit = 150 mL of wine, 360 mL of beer, or 45 mL of 40% alcohol]) or positive alcohol breath test at screening.
* Use of soft drugs (such as marijuana) within 3 months prior to the screening visit or hard drugs (such as cocaine, phencyclidine, and crack) within 1 year prior to the screening visit or positive urine drug screen at screening.
* History of allergic reactions to donepezil, piperidine derivatives, or other related drugs.
* Use of any drugs known to induce of inhibit hepatic drug metabolism (example of inducers: barbiturates, carbamazepine, phenytoin, glucocorticoids, omeprazole; examples of inhibitors: antidepressants, cimetidine, diltiazem, macrolides, imidazoles, neuroleptics, verapamil, fluoroquinolones, antihistamines) within 30 days prior to the administration of the study medications.
* Use of an investigational drug or participation in an investigational study within 30 days prior to dosing.
* Clinically significant history or presence of any gastrointestinal pathology (e.g. chronic diarrhea, inflammatory bowel diseases), unresolved gastrointestinal symptoms (e.g. diarrhea, vomiting), liver or kidney disease, or other conditions known to interfere with the absorption, distribution, metabolism, or excretion of the drug.
* Any clinically significant history or presence of neurological, endocrinal, cardiovascular, pulmonary, hematological, immunologic, psychiatric, or metabolic disease.
* Use of prescription medication within 14 days prior to administration of study medication or over-the-counter products (including natural food supplements, vitamins, or garlic as a supplement) within 7 days prior to administration of study medication, except for topical products without systemic absorption and hormonal contraceptives.
* Difficulty to swallow study medication.
* Use of tobacco products in the 3 months preceding the screening visit.
* Any food allergy, intolerance, restriction, or special diet that, in the opinion of the Medical Sub-Investigator, could contraindicate the subject's participation in this study.
* A depot injection or implant of any drug (other than hormonal contraceptives) within 3 months prior to administration of the study medication.
* Donation of plasma (500 mL) within 7 days prior to drug administration. Donation or loss of whole blood (excluding the volume of blood that will be drawn during the screening procedures of this study) prior to administration of the study medication as follows: 50 mL to 499 mL of whole blood within 30 days, or more than 499 mL of whole blood within 56 days prior to drug administration.
* Positive urine pregnancy test at screening.
* Breast-feeding subject.
* Female subjects of childbearing potential having unprotected sexual intercourse with any non-sterile male partner (i.e. male who has not been sterilized by vasectomy for at least 6 months) within 14 days prior to study drug administration.
* History of asthma or obstructive pulmonary disease.
* History of ulcer disease.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2007-06; Primary Completion 2007-07 (Actual); Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
Cmax of Donepezil. | Blood samples collected over a 72 hour period.
  Bioequivalence based on Donepezil Cmax (maximum observed concentration of drug substance in plasma).
AUC0-72 of Donepezil. | Blood samples collected over a 72 hour period.
  Bioequivalence based on Donepezil AUC0-72 (area under the concentration-time curve from time zero to time of last measurable concentration).

CONTACTS AND LOCATIONS:
Overall Officials: Benoit J Deschamps, M.D., Principal Investigator — Anapharm
Locations (1):
- Anapharm, Montreal, Quebec, Canada